CLINICAL TRIAL: NCT06820814
Title: The Association Between Physical Symptoms and Depression Among Medical Students in Egypt
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Eldaly, Director of Scientific Committee, Cairo University
Other Study IDs: Not Yet
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Depression Anxiety Disorder; Physical Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To examine the association between depression and physical symptoms among medical students in Egypt.

DETAILED DESCRIPTION:
The Google Form will be open for one week from the start of the academic term. It is divided into three parts:

Demographic Data - which includes age, academic level, relationship status, and whether the student intends to work while studying.

Patient Health Questionnaire PHQ-9: Assesses symptoms of poor mental health in the two weeks prior to the start of term.

Patient Health Questionnaire PHQ-15: This is a measure of physical symptoms felt in the week prior to the commencement of the academic term.

The questionnaire will be distributed among different medical faculties in Egypt and all students will be required to fill it out. Data analysis will be done through SPSS to explore the relationship between psychological and physical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Medical students enrolled in any medical program in Egypt.
* Age range: Typically 19 to 30 years (or based on your study's demographic focus).
* Willingness to participate and provide informed consent.
* Self-reported symptoms of depression: Those who indicate moderate to severe symptoms on screening tools (e.g., PHQ-9).
* Physical symptoms: Those who report experiencing physical symptoms (e.g., headaches, fatigue, gastrointestinal discomfort, etc.) on a checklist.

Exclusion Criteria:

* Non-medical students (students outside of the medical program).
* Students with a history of major medical conditions that may confound the physical symptoms (e.g., chronic diseases like diabetes, hypertension, or neurological disorders).
* Students with a diagnosed psychiatric disorder (e.g., bipolar disorder, schizophrenia, etc.) or those already undergoing psychiatric treatment.
* Non-consenting individuals: Students who decline to participate in the study or do not provide informed consent.
* Incomplete responses: Students who fail to provide adequate or valid responses in the questionnaires.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Medical students enrolled in any medical program in Egypt.
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
PATIENT HEALTH QUESTIONNAIRE (PHQ-9) | 1 week
  The Patient Health Questionnaire-9 (PHQ-9) used for screening, diagnosing, monitoring, and measuring the severity of depression.
  It consists of nine questions; Each item is scored from 0 (Not at all) to 3 (Nearly every day), leading to a total score ranging from 0 to 27.
  Scores can be categorized as follows:
  1-4: Minimal or no depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression
PATIENT HEALTH QUESTIONNAIRE PHYSICAL SYMPTOMS (PHQ-15) | 1 week
  PATIENT HEALTH QUESTIONNAIRE PHYSICAL SYMPTOMS (PHQ-15) used to assess the severity of somatic (physical) symptoms.
  Consists of 15 common physical symptoms (e.g., stomach pain, dizziness, fatigue).
  Each symptom is rated based on how much it has bothered the individual in the past 7 days.
  Scoring system:
  0 = Not bothered at all
  1. = Bothered a little
  2. = Bothered a lot Total score range: 0 to 30 Minimal: 0-4 Low: 5-9 Medium: 10-14 High: 15-30

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt